CLINICAL TRIAL: NCT06162481
Title: Admission Time and Outcomes of Patients Admitted to Intensive Care Unit in a Tertiary Level Teaching Hospital
Status: Completed | Type: Observational
Sponsor: Tribhuvan University Teaching Hospital, Institute Of Medicine. (Other)
Responsible Party: Principal Investigator, Ashmita Paudel, Principal Investigator, Tribhuvan University Teaching Hospital, Institute Of Medicine.
Other Study IDs: 4 4 2 ( 6 - 1 1 ) 6 2
Record Dates: First submitted 2023-11-22; First posted 2023-12-08 (Actual); Last update posted 2023-12-08 (Actual); Status verified 2023-11

CONDITIONS: FOCUS of Study: Time of Admission to ICU and Outcome

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Admitted during office hours
- Admitted off hours

SUMMARY:
An intensive care unit (ICU) is a specialized unit within the hospital where patients who need immediate medical attention are admitted both during office hours and off hours.1 Literatures report reduced working efficiency because of long working hours, unavailability of 24/7 intensivist staffing and the absence of the same level of hospital services like laboratory investigations during off hours affecting outcome of the patients. 2-6 High intensity staffing model and shorter workhours can improve the outcome.7 However, these are not always feasible in ICUs of low and middle income countries like Nepal. Any variations in outcome depending upon time of ICU admission may impact the workforce planning, medical insurance, and healthcare policy.

The aim of this study was to compare the outcomes of patients admitted to the ICU during office hours and off hours in terms of ICU mortality, duration of mechanical ventilation and length of stay.

ELIGIBILITY:
Inclusion Criteria:

- age >= 16 years

Exclusion Criteria:

* Patient who were discharged on request, left against medical advice, had withdrawal of active life support

Min Age: 16 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: All patients admitted to ICU
Sampling Method: Non-Probability Sample
Enrollment: 3242 (Actual)
Dates: Start 2023-03-15 (Actual); Primary Completion 2023-08-31 (Actual); Study Completion 2023-08-31 (Actual)

PRIMARY OUTCOMES:
ICU length of stay | Each patient will be followed till death or discharge alive from ICU whichever occurs earlier
days of mechanical ventilation | Each patient will be followed till death or liberation from Mechanical ventilation whichever occurs earlier
In ICU mortality | each patient will be followed till death or discharge from ICU whichever is earlier

CONTACTS AND LOCATIONS:
Locations (1):
- Tribhuvan University Teaching Hospital, Kathmandu, Bagmati, Nepal

IPD SHARING:
Plan to Share IPD: No